CLINICAL TRIAL: NCT02378064
Title: Comparison of Fimasartan Versus Amlodipine Therapy on Carotid PlaquE Inflammation
Acronym: FACE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CHEOL WHAN LEE, M.D., Ph.D (Other)
Collaborators: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor-Investigator, CHEOL WHAN LEE, M.D., Ph.D, professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: AMCCV2014-10
Record Dates: First submitted 2015-02-26; First posted 2015-03-04 (Estimated); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Inflammation Plaque, Atherosclerotic; Coronary Disease; Renin-Angiotensin System
Keywords: Fluorodeoxyglucose F18; Positron-Emission Tomography and Computed Tomography; Plaque, Atherosclerotic; Renin-Angiotensin System
MeSH Terms: conditions — Coronary Disease; Plaque, Atherosclerotic | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Fimasartan and vytorin (Experimental): fimasartan(60mg,QD)+Vytorin(10mg,QD)
  Interventions: Drug: 6-month treatment
- Fimasartan and rosuvastatin (Experimental): fimasartan(60mg,QD)+rosuvastatin(5mg,QD)
  Interventions: Drug: 6-month treatment
- amlodipine and vytorin (Active Comparator): amlodipine(5mg,QD)+Vytorin(10mg,QD)
  Interventions: Drug: 6-month treatment
- amlodipine and rosuvastatin (Active Comparator): amlodipine(5mg,QD+rosuvastatin(5mg,QD)
  Interventions: Drug: 6-month treatment

INTERVENTIONS:
Drug: 6-month treatment

SUMMARY:
The purpose of this study is to evaluate the effects of angiotensin receptor 1 blocker versus calcium channel blocker on atherosclerotic plaque inflammation using serial FDG PET/CT imaging of carotid artery.

ELIGIBILITY:
Inclusion Criteria:

* Men or Women at least 18 years of age inclusive
* Patients with acute coronary syndromes or unstable angina pectoris
* Hypertension or blood pressure more than 140/90mmHg
* FDG PET/CT shows at least 1 hot uptakes at carotid and or ascending aorta
* The patient or guardian agrees to the study protocol and the schedule of clinical and FDG PET/CT follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethical Committee of the respective clinical site.

Exclusion Criteria:

* Patients treated with carotid endarterectomy or stent placement
* Chronic disease requiring treatment with oral, intravenous, or intra-articular corticosteroids (use of topical, inhaled, or nasal corticosteroids is permissible).
* Untreated hyperthyroidism, or hypothyroidism
* Any clinically significant abnormality identified at the screening visit, physical examination, laboratory tests, or electrocardiogram which, in the judgment of the Investigator, would preclude safe completion of the study.
* Evidence of congestive heart failure, or left ventricular ejection fraction < 40%.
* Significant renal disease manifested by serum creatinine > 2.0mg/dL, or creatinine clearance of < 40 ml/min (by Cockcroft-Gault method).
* Hepatic disease or biliary tract obstruction, or significant hepatic enzyme elevation (ALT or AST > 3 times upper limit of normal).
* History of adult asthma manifested by bronchospasm in the past 6 months, or currently taking regular anti-asthmatic medication(s).
* Unwillingness or inability to comply with the procedures described in this protocol.
* Patient's pregnant or breast-feeding or child-bearing potential.
* Type I Diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-05; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
change (follow-up minus baseline) in standardized FDG uptake value | 6month
  change (follow-up minus baseline) in standardized FDG uptake value within the regions of interest, known as a target-to-background ratio (blood-normalized standardized uptake value).

SECONDARY OUTCOMES:
changes of blood pressure | 6month
  systolic and diastolic
Serial changes of lipid battery | 6month
  total cholesterol, triglyceride, HDL-cholesterol, LDL-cholesterol

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Oh M, Kim H, Shin EW, Sung C, Kim DH, Moon DH, Lee CW. Effects of ezetimibe/simvastatin 10/10 mg versus Rosuvastatin 10 mg on carotid atherosclerotic plaque inflammation. BMC Cardiovasc Disord. 2019 Aug 19;19(1):201. doi: 10.1186/s12872-019-1184-2. PMID 31426749